CLINICAL TRIAL: NCT00343070
Title: Functional Neuroimaging in Depression: Longitudinal Study of PET Metabolism in Correlation With Changes in Attentional Bias, Autobiographical Memory, Future Fluency and Facial Recognition in Depressed Patients Treated With Escitalopram.
Brief Title: Functional Neuroimaging in Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); H. Lundbeck A/S (Industry)
Responsible Party: Kurt Audenaert, University Hospital Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/176
Record Dates: First submitted 2006-06-19; First posted 2006-06-22 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oral administration of escitalopram during 8 weeks

SUMMARY:
Oral administration of escitalopram during 8 weeks; PET scan with 18F-FDG at inclusion and after 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Major Depression, Depressive episode, following DSM-IV criteria
* MADRS-score > 25
* Age: 18-65 yrs
* Medication-free or anti-depressant wash-out 7 days (for fluoxetine: 6 weeks)
* Lorazepam 1mg or zolpidem 10mg are allowed

Exclusion Criteria:

* Suicidality
* Bipolar disorder, following DSM-IV criteria
* Psychotic symptoms
* Substance abuse
* Personality disorder, following DSM-IV criteria
* Cognitive dysfunction due to trauma capitis or dementia
* Diabetes mellitus
* Women without contraceptive protection, with pregnancy or breast feeding
* Pharmacological treatment or ingestion of substance that can influence cerebral perfusion less than a month before inclusion
* IQ below 80
* Conditions not compatible with SPC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Brain metabolism

SECONDARY OUTCOMES:
Cognitive functions
Efficacy scales (mood, anxiety, anger and hopelessness)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Audenaert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - University Hospital Ghent, Ghent
  - AZ Groeninge campus Sint Maarten, Kortrijk

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be